CLINICAL TRIAL: NCT01667666
Title: A Clinical Study to Determine if Nebulized Hypertonic Saline Attenuates Acute Lung Injury Following Trauma and Hemorrhagic Shock
Brief Title: Clinical Trial of Nebulized Hypertonic Saline to Attenuate Post-Traumatic Acute Lung Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low enrollment and loss of funding
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Professor of Surgery, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COMIRB #11-0706
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Acute Lung Injury; Adult Respiratory Distress Syndrome
Keywords: trauma; acute lung injury; adult respiratory distress syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nebulized HTS (Experimental): The first 5 patients will receive 3% Nebulized hypertonic saline, the second 5 patients will receive 4.5% Nebulized hypertonic saline, the third group 6% Nebulized hypertonic saline, and the fourth group of 5 patients will receive 7% Nebulized hypertonic saline. The nebulizer is dosed 2-3 times a day for 36 hours.
  Interventions: Drug: Nebulized hypertonic saline

INTERVENTIONS:
Drug: Nebulized hypertonic saline — The first 5 patients will receive 3% hypertonic saline in a nebulizer, the second 5 patients will receive 4.5% nebulized hypertonic saline, the third group 6% nebulized hypertonic saline, and the fourth group of 5 patients will receive 7% nebulized hypertonic saline. The nebulizer is dosed 2-3 times a day for 36 hours.

SUMMARY:
This study evaluates the use of nebulized hypertonic saline (aerosolized salt water) as a preventive treatment for post-traumatic acute lung injury (ALI). Both animal and human research indicate that aerosolized salt water might help reduce harmful inflammation with minimal risks.

DETAILED DESCRIPTION:
Despite over 40 years of investigation, acute lung injury (ALI) remains a leading cause of morbidity in critically ill patients, and a disease for which there is no effective pharmacologic therapy. Our group and others have focused on the anti-inflammatory effects of intravenous hypertonic saline (HTS) acting on the injured endothelium with promising results experimentally, but failed to confirm the benefit clinically. Recent work, however, has shown that inhaled or nebulized HTS targeted at the epithelium is safe and effective in treating cystic fibrosis, COPD, and neonatal bronchiolitis. Recognizing the central role of the pulmonary epithelium in ALI, nebulization has the advantage of achieving high concentrations of the therapy without producing systemic side effects. Thus, we hypothesize that nebulized hypertonic saline will attenuate acute lung injury following trauma.

ELIGIBILITY:
Inclusion Criteria:

* adult 18 ≤ age ≤ 65
* trauma with a 9 ≤ NISS ≤ 36
* ≤10 units of RBC in the first 6 hours (as this is a major risk factor for ARDS and MOF in this population)

Exclusion Criteria:

* Direct or indirect lung injury
* Elevated intracranial pressure requiring treatment, including but not limited to mannitol, intravenous hypertonic saline, and ventricular drainage
* History of severe chronic respiratory disease
* Child-Pugh Class C liver failure
* Prisoners
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
change in the respiratory parameters | baseline and every 6 hours for 36 hours
  For intubated patients - A decrease greater than 20% in PaO2/FiO2 (P/F) ratios will trigger DSMB review. For not intubated patients - a) the need to increase FiO2 by 10% (approximate 4 liter/minute increase) to maintain a peripheral oxygen saturation (SaO2) of 90% during nebulizer treatment; b) evidence of respiratory distress (as documented in the chart by the patient's attending) during nebulizer treatment; and c) respiratory insufficiency requiring intubation and mechanical ventilation at any point will trigger DSMB review.

SECONDARY OUTCOMES:
death within 28 days | 28 days or discharge
  If the rate of death within 28 days for this patient population is less than 50% the expected rate for every 5 patients based on our clinical trauma database over the past 5 years, a DSMB review will be triggered.
lung dysfunction scores | baseline and 28 days or discharge
  Denver lung MOF score will be measure daily until discharge or 28 days, which ever is first. For every 5 patients, if the rate of lung dysfunction for this patient population is less than 50% the expected rate based on our clinical trauma database over the past 5 years, a DSMB review will be triggered.
ventilator-free days (VFD) | baseline and 28 days or discharge
  Ventilator free days will be tracked with 28 days as a reference. If the number of VFDs for this patient population is greater than one standard deviation of the predicted value for every 5 patients based on our clinical trauma database over the past 5 years, a DSMB review will be triggered.
MOF scores (Denver MOF score) | 28 days or discharge
  Denver MOF score will be recorded daily until discharge or 28 days, which ever is sooner. for every 5 patients, if the rate of MOF for this patient population is greater than one standard deviation of the predicted value for every 5 patients based on our clinical trauma database over the past 5 years, a DSMB review will be triggered

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E Moore, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States